CLINICAL TRIAL: NCT02371109
Title: SYSTEMATIC: NAATS of Pooled Selftaken Versus Clinicantaken Swabs 1
Status: Completed | Type: Observational
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: GU12/10329
Record Dates: First submitted 2015-01-26; First posted 2015-02-25 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- selftaken vs clinical taken swabs
  Interventions: Other: selftaken versus clinically taken swabs

INTERVENTIONS:
Other: selftaken versus clinically taken swabs

SUMMARY:
Routine screening for gonorrhoea and chlamydia involves urine samples in males and selftaken vulvovaginal swabs (VVSs) in females. As well as infecting the urethra (pee tube) and cervix (neck of womb), gonorrhoea and chlamydia may also infect the rectum (bottom) and throat (both called extragenital sites), often with no symptoms. In some people infection will be found at more than one site, but in others it will only be in one, and if all anatomical sites are not tested some infections will be missed. In certain women one third of infections may be missed, in men who have sex with men (MSM) up to 90% may be missed, if extragenital swabs are not taken. Currently, routine community testing does not include extragenital sites. Until recently these samples could not easily be taken outside clinical settings (hospitals, clinics or surgeries), but new DNA tests for gonorrhoea, called NAATs, now make this possible.

However, they are expensive, and taking samples from extragenital sites would treble the costs. We propose that swabs from the three sites per person are pooled and analysed together rather than tested separately. This method would identify whether the person had the infection but not the anatomical site; this would not alter the management of the individual. Swabs from the rectum and throat have historically been taken by clinicians (doctors or nurses). The main attraction of community screening is that it is client led using selftaken samples. Recent studies suggest that selftaken swabs from the rectum and throat are acceptable to clients and may be as good as swabs taken by clinicians, but the costeffectiveness of this approach has not been investigated. Our aim is to establish whether in MSM and females selftaken samples that are pooled and processed by NAATs are as effective as the individual tests taken by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Attending the Leeds Centre for Sexual Health for an appointment where diagnostic tests for gonorrhoea and chlamydia will be taken Aged 16 or over

Exclusion Criteria:

* Attending the Leeds Centre for Sexual Health for an appointment where diagnostic tests for gonorrhoea and chlamydia will be taken Aged 16 or over

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is all patients who attend the Leeds Centre for Sexual Health for an appointment where diagnostic tests for gonorrhoea and chlamydia. All will be given the opportunity to take part in the research project.
Sampling Method: Probability Sample
Enrollment: 1786 (Actual)
Dates: Start 2014-12-09 (Actual); Primary Completion 2016-09-19 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of the self taken swabs analysed together as a pooled sample, compared with individually analysed (nonpooled) clinican taken samples. | The study duration

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

REFERENCES:
- [Derived] Wilson JD, Wallace HE, Loftus-Keeling M, Ward H, Davies B, Vargas-Palacios A, Hulme C, Wilcox MH. Swab-Yourself Trial With Economic Monitoring and Testing for Infections Collectively (SYSTEMATIC): Part 2. A Diagnostic Accuracy and Cost-effectiveness Study Comparing Rectal, Pharyngeal, and Urogenital Samples Analyzed Individually, Versus as a Pooled Specimen, for the Diagnosis of Gonorrhea and Chlamydia. Clin Infect Dis. 2021 Nov 2;73(9):e3183-e3193. doi: 10.1093/cid/ciaa1546. PMID 33044490
- [Derived] Wilson JD, Wallace HE, Loftus-Keeling M, Ward H, Davies B, Vargas-Palacios A, Hulme C, Wilcox MH. Swab-yourself Trial With Economic Monitoring and Testing for Infections Collectively (SYSTEMATIC): Part 1. A Diagnostic Accuracy and Cost-effectiveness Study Comparing Clinician-taken vs Self-taken Rectal and Pharyngeal Samples for the Diagnosis of Gonorrhea and Chlamydia. Clin Infect Dis. 2021 Nov 2;73(9):e3172-e3180. doi: 10.1093/cid/ciaa1266. PMID 32877521